CLINICAL TRIAL: NCT06008626
Title: Multicenter Pilot Study of the Cryosa System for the Treatment of Obstructive Sleep Apnea
Brief Title: Clinical Trial of the Cryosa System for the Treatment of Obstructive Sleep Apnea
Acronym: ARCTIC-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cryosa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11515
Record Dates: First submitted 2023-08-07; First posted 2023-08-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cryosa Procedure (Experimental): The purpose of this study is to evaluate the safety and effectiveness of Cryosa System applied to the tongue and soft palate in patients with clinically diagnosed obstructive sleep apnea (OSA).
  Interventions: Device: Cryosa Procedure

INTERVENTIONS:
Device: Cryosa Procedure — Cryotherapy
  Other Names: OSA Cryotreatment

SUMMARY:
This is a prospective, multicenter, non-randomized single-arm safety and performance study to collect data to evaluate the safety of the Cryosa procedure to treat obstructive sleep apnea (OSA) in patients with moderate to severe OSA. The study will also evaluate the chronic performance of the Cryosa system and collect clinical measures for therapy effectiveness that will be used to demonstrate safety and effectiveness in the next clinical study.

DETAILED DESCRIPTION:
The study will treat 25 subjects enrolled at up to 10 sites in the United States. Enrollment is competitive but each site will be limited to 15 subjects treated.

ELIGIBILITY:
Inclusion Criteria:

1. To participate in this study, the subject must meet ALL of the following inclusion criteria:
2. Age 22 - 70 years
3. Not able to use, refuse to use or intolerant of Positive Airway Pressure (PAP) or Mandibular Advancement Device (MAD) if using, must be < 4 hours per night, < 5 days/week.
4. Failed, are not candidates for, or have refused other invasive procedures such as hypoglossal nerve stimulation or pharmacotherapy for the primary treatment of OSA such as Tirzepatide.
5. BMI ≥30 or ≤ 40 kg/m2 at enrollment
6. AHI ≥30 at enrollment based on in-lab polysomnography study OR AHI ≥ 15 and BMI of ≥ 30 at enrollment based on in-lab polysomnography study Is geographically stable and in close proximity to the site
7. Able and willing to provide written consent to participate in the study

Exclusion Criteria:

1. Contraindication to general anesthesia or in the opinion of the Investigator would not be able to tolerate the procedure, including intubation during the procedure or in response to an adverse event
2. Actively taking ACEs/ARBs
3. Actively undergoing immunotherapy (Allergy shots)*, or unwilling to washout of allergy shots at least 2 weeks prior to study procedure.

   * Patients receiving immunotherapy may be eligible if they undergo a 2-week wash-out prior to the study procedure
4. Severe uncontrolled asthma
5. Severe maxillary mandibular insufficiency that in the opinion of the investigator thought to be the primary cause of OSA
6. Obvious severe fixed upper airway obstructions (tumors, polyps, nasal obstruction)
7. Previous surgery within 12 weeks of scheduled procedure performed on the soft tissue of the upper airway (e.g., uvula, soft palate, or tonsils).
8. Oral cancer or non-healing oral wounds
9. Prior sleep surgeries, including tongue base reduction, UPPP and hypoglossal nerve stimulation.
10. History of radiation therapy to neck or upper respiratory tract
11. Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat (with exception of tonsillectomy and/or adenoidectomy)
12. History presence of cold urticaria at the time of screening History of cryoglobulinemia
13. History of allergy to glycerin
14. History of hospitalization with mechanical ventilation due to COVID-19 per investigator discretion
15. Resistant hypertension defined as a blood pressure that remains above goal despite concurrent use of three antihypertensive agents of different classes taken at maximally tolerated doses
16. Patients with diagnosed autoimmune disorders including thyroid disease, lupus, multiple myeloma, chronic lymphocytic leukemia
17. Neuromuscular disease or other neurologic deficits (for example multiple sclerosis, muscular dystrophy, Parkinson's disease, transient ischemic attack, epilepsy or cerebrovascular accident)
18. Diagnosis of any moderate to severe congestive obstructive pulmonary disease (COPD)
19. Active, severe pulmonary vascular disease (for example pulmonary arterial hypertension or pulmonary embolism) History of angioedema of the airway
20. Hereditary angioedema and other autoimmune disorders that could lead to acquired angioedema - confirmed with a compliment component C4 blood test <13mg/dL.
21. Uncontrolled Diabetes (including Diabetes Mellitus [DM] or Insulin Dependent Diabetes Mellitus [IDDM]) with HbA1c >9.
22. Currently receiving treatment for severe cardiac valvular dysfunction, NYHA Class III or IV heart failure, unstable angina or recent (< 12 months) myocardial infarction or severe cardiac arrhythmias
23. Subjects with bleeding event, known bleeding diathesis, impaired immunity for any reason, or heart attack or stroke within the last 12 months
24. Clinical evidence of severe renal failure (Stage 4 or 5) undergoing dialysis or expected to institute dialysis within 6 months
25. History or current clinical evidence of TIA or stroke or muscular dysfunction
26. Current smoker (≥ 1 pack/day)
27. Presence of occupational shift work or anticipation of shift changes during the next 2 years
28. Subject has sleep hygiene behavior that is likely to interfere with measurement outcomes during PSG and/or HSAT
29. Known active substance use disorder
30. Other severe sleep disorders that in the opinion of the investigator, confound functional assessments of sleepiness such as narcolepsy with cataplexy, severe insomnia/insomnia secondary to chronic pain, PTSD
31. Patients taking any of the following medication that could affect study endpoints: benzodiazepines, Z-drugs (zolpidem and eszopiclone) opiates, antipsychotics (neuroleptics), phenothiazines, and prescription stimulants (including Sunosi, Provigil, and Nuvigil)
32. Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject's ability to meet study requirements and ability to provide study consent
33. Females who are pregnant or females of childbearing age with intention to become pregnant during the study period (≤ 3 months from treatment date)
34. Any other reason the investigator deems subject is unfit for participation in the study
35. Subject currently participating in other premarket investigational studies unless approved by Sponsor in writing

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Procedure or Device/ Treatment Related Events | First 90 days post-procedure
  Safety will be assessed by evaluating all serious procedure- or device/treatment-related events occurring in the first 90 days post-procedure.
  Adverse events (AE), both serious and non-serious, related and unrelated, will be collected from all subjects enrolled for the duration of the study.

SECONDARY OUTCOMES:
Sleep Testing | 6 Month Follow-up Visit
  Quantify the effect of the Cryosa procedure in reducing the severity of OSA post-procedure by evaluating the change from baseline in the apnea hypopnea index (AHI4) with polysomnography (PSG) testing.
Patient Reported Outcomes (PRO) Efficacy Measures - Epworth Sleepiness Survey (ESS) | 30 Days, 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Evaluate change in daytime sleepiness after treatment compared to baseline.
Patient Reported Outcomes (PRO) Safety Measures - Pain Numeric Scale (NRS) | 7 Days, 30 Days, 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Evaluate oropharyngeal pain metrics after treatment compared to baseline.
Patient Reported Outcomes (PRO) Safety Measures - Eating Assessment Tool (EAT-10) | 7 Days, 30 Days, 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Evaluate change in swallowing metrics after treatment compared to baseline.
Patient Reported Outcomes (PRO) Safety Measures - PROMIS-Sleep Disturbance (PROMIS-SD) | 30 Days, 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Assess perception of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness
Patient Reported Outcomes (PRO) Safety Measures - PROMIS-Sleep Related Impairment (PROMIS-SRI) | 30 Days, 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Assess a range of symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles

OTHER OUTCOMES:
Home Sleep Apnea Testing (HSAT) - Apnea-Hypopnea Index (AHI4) | 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Two nights of testing will be collected, and the average of the two nights will be used to evaluate the change in AHI4 after treatment compared to baseline.
Home Sleep Apnea Testing (HSAT) - Oxygen Desaturation Index (ODI) | 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Two nights of testing will be collected, and the average of the two nights will be used to evaluate the change in ODI sleep metrics after treatment compared to baseline.
Home Sleep Apnea Testing (HSAT) - Oxygen Saturation (SpO2) | 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Two nights of testing will be collected, and the average of the two nights will be used to evaluate the change in SpO2 sleep metrics after treatment compared to baseline.
Home Sleep Apnea Testing (HSAT) - Hypoxic Burden | 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Two nights of testing will be collected, and the average of the two nights will be used to evaluate the change in hypoxic burden sleep metrics after treatment compared to baseline.
Home Sleep Apnea Testing (HSAT) - Snoring | 90 Days, 6 Months, 12 Months, 18 Months and 24 Months Post-procedure
  Two nights of testing will be collected, and the average of the two nights will be used to evaluate the change in snoring episodes sleep metrics after treatment compared to baseline.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UCHealth University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Albany ENT & Allergy Services, Albany, New York
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Tennessee Health Sciences Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No